CLINICAL TRIAL: NCT06126328
Title: EASE Study: A Randomized, Controlled Study to EvAluate the Safety and Effectiveness of the Materna Prep Device to Pre-stretch the Vaginal Canal and Pelvic Floor Muscles in Preparation for Vaginal Delivery
Brief Title: Materna Prep Study Phase II
Acronym: EASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Materna Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CP0001.G
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Vaginal Delivery; Pelvic Organ Prolapse
Keywords: Pelvic Floor Health; Levator Ani Muscle Injury; Pelvic Floor Injury; Vaginal Delivery; Childbirth; Complications
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: Ultrasound images are assessed by physicians blinded to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Materna Prep Device (Active Comparator): Materna Prep Device
  Interventions: Device: Materna Prep Device
- Standard of Care (SOC) (No Intervention): Standard of Care Control

INTERVENTIONS:
Device: Materna Prep Device — Subjects are treated with Materna Prep Device prior to vaginal delivery
  Arms: Materna Prep Device

SUMMARY:
This study is designed to evaluate the safety and effectiveness of the Materna Prep Device in reducing pelvic muscle injuries during vaginal delivery.

Subjects are randomized to Materna Prep Device or Standard of Care without use of the Materna Prep Device

Intervention with the Materna Prep Device is expected to be a one-time use of approximately 30-90 minutes during the 1st stage of labor.

Subject participation in the study is targeted to be 3 months from the time of the use of the device during delivery with optional long-term follow-up.

DETAILED DESCRIPTION:
Vaginal delivery is a major risk factor for pelvic floor dysfunction. Clinical aspects of pelvic floor dysfunction include pelvic organ prolapse, sexual dysfunction, and fecal and urinary incontinence. Trauma to the pelvic structures occurs as the fetal head passes through the vaginal canal, especially with acute distension at the time of crowning - the exiting of the fetal head.

The Materna Prep Device is a single-use, semi-automated dilator used during the first phase of labor in order to prepare the vaginal canal for vaginal delivery. By slowly pre-stretching the vagina and surrounding pelvic tissues during labor, the device is essentially dictating the strain rate of the tissue during labor. In previous feasibility studies, the elastic recovery of the tissue has been shown to be on the order of several hours, allowing the benefits of pre-stretching the vagina and surrounding pelvic tissues to last throughout labor. The device is intended to be removed prior to the initiation of the second stage of labor, for delivery to occur unobstructed.

The target patient population for this study is nulliparous women entering the first phase of labor and scheduled for vaginal delivery with an epidural.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled for vaginal birth.
2. Subject is gestating a single fetus.
3. Subject is nulliparous, or had a previous pregnancy terminated within 24 weeks gestation.
4. Subject is able and willing to comply with the protocol required follow-up visits.
5. Subject is able and willing to provide written informed consent prior to enrollment.
6. In the opinion of the Investigator, the subject has sufficient mental capacity to understand the informed consent form (ICF), comply with the protocol requirements, and provide clinically relevant and reliable feedback regarding their experience with the device.
7. Subject receives epidural anesthesia during labor prior to enrollment.
8. Subject is 18 years of age or older at time of consent.

Exclusion Criteria:

1. Subject has high likelihood of less than 1 hour of potential device dilation time after she arrives at the hospital.
2. Subject is planning or requires a Caesarean-section prior to randomization.
3. Subject begins labor with less than 36 weeks gestation.
4. Subject has a neurological disorder that could cause pelvic floor dysfunction, such as multiple sclerosis or spinal cord injury.
5. Subject has a collagen-associated disorder that affects tissue elasticity, such as scleroderma or Ehlers-Danlos syndrome.
6. Subject has a localized (genital tract) or systemic infection.
7. Subject has a medical history which could lead to pelvic floor dysfunction, such as prior pelvic fractures, pelvic soft tissue injuries, or vaginal surgery.
8. Subject has any general health condition or systemic disease that may represent, in the opinion of the Investigator, a potential increased risk associated with device use or pregnancy.
9. Subject has placenta previa or vasa previa.
10. Subject has known significant chromosomal or structural fetal anomalies.
11. Subject has a category 2 and/or 3 fetal tracing that is unresolved.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 214 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The occurrence of pelvic muscle injury, defined as complete or partial detachment of the levator ani muscle diagnosed via ultrasound imagingmuscle diagnosed via ultrasound imaging | 3-month Follow-up
  Use transperineal ultrasound to identify levator ani muscle detachment

SECONDARY OUTCOMES:
The occurrence of pelvic muscle injury, defined as complete detachment of the levator ani muscle diagnosed via ultrasound imaging | 3-month Follow-up
  Use transperineal ultrasound to identify levator ani muscle detachment
Length of 2nd Stage Labor | Day of Delivery
  Compare the length of the second stage of labor, defined as the time from the cervix being dilated to 10 cm to the complete delivery of the baby between study groups.
Levator Hiatal Area | 3-month Follow-up
  Compare the levator hiatal area (cm2 - measurement between pelvic muscle and pelvic bone)
Perineal Lacerations | Day of Delivery
  Compare the rate of perineal lacerations determined by visual insepction post-delivery between study groups
Obstetric anal sphincter injury - OASI | Day of Delivery
  Compare the rate of tearing of the muscles of the anal sphincter between study groups.
Obstetric anal sphincter injury - OASI | 3-month Follow-up
  Compare the rate of tearing of the muscles of the anal sphincter on ultrasound between study groups.
C-Sections | Day of Delivery
  Compare the rate of C-Section due to arrest of labot in the second stage
Infant APGAR scores | Day of Delivery
  Compare infant APGAR scores between study groups.
Qualitative pelvic health feedback | 3-month Follow-up
  Compare qualitative pelvic health feedback assessed by PFIQ-7and PFDI-20 Questionnaires
Operative Delivery | Day of Delivery
  Compare the rate of instrument use in vaginal deliveries between study groups
First Push to Delivery | Day of Delivery
  Compare the mean time form first push to delivery between study groups.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Christiana Care - Center for Women's & Children's Health, Newark, Delaware
  - Mayo Clinic, Rochester, Minnesota
  - The Cooper Health System, Camden, New Jersey
  - Rutgers Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - The Metro Health System, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Lewis Katz School of Medicine at Temple, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No